CLINICAL TRIAL: NCT06950606
Title: Pneumatic Leg Compression and Norepinephrine Requirements in Patients Having Non-cardiac Surgery: a Pilot Monocentric Prospective Randomized Interventional Clinical Trial
Brief Title: Pneumatic Leg Compression and Norepinephrine Requirements in Patients Having Non-cardiac Surgery
Acronym: PLANE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-101383-BO-ff
Record Dates: First submitted 2025-04-21; First posted 2025-04-30 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Hypotension During Surgery
Keywords: Stressed volume; Vasopressor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pneumatic leg compression (Experimental): PLC group (i.e., intervention group):
  Patients assigned to the PLC group will receive a pneumatic lower limb compression sleeve during surgery.
  Interventions: Device: Pneumatic leg compression
- Routine care (No Intervention): Routine care group (i.e., control group):
  Patients assigned to the Routine care group will not receive a pneumatic lower limb compression sleeve. There will be no standardized anesthesia management protocol; all decisions regarding hemodynamic management will be made at the discretion of the treating anesthesiologist.

INTERVENTIONS:
Device: Pneumatic leg compression — Patients assigned to the PLC group will receive a pneumatic leg compression sleeve encompassing the calf and thigh, with sleeve size adjusted according to thigh circumference and manufacturer recommendations. The compression pump will be activated before the start of surgery. After surgery, the responsible trial personnel will deactivate the pump and remove the compression sleeves in the PLC group. There will be no standardized anesthesia management protocol; all decisions regarding hemodynamic management will be made at the discretion of the treating anesthesiologist
  Arms: Pneumatic leg compression

SUMMARY:
The PLANE trial is a randomized, single-center trial investigating whether pneumatic leg compression reduces the amount of norepinephrine needed to keep MAP above 65mmHg compared to routine care without PLC in patients having non-cardiac surgery under general anesthesia

ELIGIBILITY:
Inclusion Criteria:

Consenting patients ≥45 years scheduled for elective non-cardiac surgery under general anesthesia that is expected to last ≥60 minutes

Exclusion Criteria:

Patients with the following exclusion criteria:

* Surgery in which pneumatic calve compression is indicated according to ERAS guidelines
* Surgery which interferes with the installation or correct function of PLC
* Sepsis (according to current Sepsis-3 definition)
* Pregnancy
* Congestive heart failure NYHA III/IV
* American Society of Anesthesiologists (ASA) physical status classification V or VI
* Interference of PLC and patient positioning (e.g.; extreme Trendelenburg positioning, lithotomy positioning)
* Contraindications for the use of PLC according to the German guideline13 (e.g., extensive thrombophlebitis, thrombosis or suspected thrombosis of the lower limbs, erysipelas, acute phlegmon, limb compartment syndrome, severe uncontrolled arterial hypertension, lymphatic drainage disorder proximal to PLC, extensive open soft tissue trauma, autoimmune blistering skin conditions such as IgA bullous dermatosis or bullous pemphigoid)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Average norepinephrine infusion rate | Intraoperative
  Average intraoperative norepinephrine infusion rate [μg kg-1 min-1] needed to keep MAP above 65mmHg. The average intraoperative norepinephrine infusion rate will be calculated using the absolute amount of norepinephrine administered per kg bodyweight [μg kg-1] divided by the duration of surgery (between surgical incision and suture) [min] (continuous outcome)

SECONDARY OUTCOMES:
Average norepinephrine infusion rate | Perioperative
  Average norepinephrine infusion rate [μg kg-1 min-1] needed to keep MAP above 65mmHg. (continuous outcome)
Amount of hypotensive events | Intraoperative
  Amount of hypotensive events with a MAP <65 [mmHg]
Lowest MAP | Intraoperative
  Lowest MAP [mmHg]
Cumulative amount of hypotensive time | Intraoperative
  Cumulative amount of hypotensive time with a MAP <65 mmHg [min]
Time-weighted average MAP <65 mmHg | Perioperative
  Time-weighted average MAP <65 mmHg (area under a MAP of 65 mmHg divided by the time from the beginning of induction of general anesthesia until the end) [mmHg]
Crystalloid fluid application | Intraoperative
  Amount of crystalloid fluid application [ml]

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No